CLINICAL TRIAL: NCT04508517
Title: A Cohort Study on the Etiology and Pathological Types of Brain White Matter Injury in Late Preterm Infants
Brief Title: Brain White Matter Injury in Late Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Dan Chen, Attending doctor，Principal Investigator, Shengjing Hospital
Other Study IDs: DChen
Record Dates: First submitted 2020-08-03; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: White Matter Injury
Keywords: white matter injury;late preterm infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
At 34 weeks, the brain weight of preterm infants is only 65% that of term infants, and the cortex volume is 53% that of term infants. Damage at this stage of development will also change the trajectory of specific processes in the development of neurons and glial cells, resulting in neurological dysfunction in survivors.The incidence of cerebral palsy in late preterm infants is three times higher than in term infants, and about 25% lag behind term infants in learning, language and other neurodevelopment. At 34-37 weeks of gestation, oligodendrocytes are still late oligodendrocyte precursors and vascular development of the white matter area is immature, making the brain more prone to white matter injury (WMI).

DETAILED DESCRIPTION:
1.1Patients Late preterm infants who were hospitalized in Shengjing Hospital from 1st January 2009 to 31st December 2022.

Risk factors prompting MRI evaluation included: (1) premature rupture of fetal membrane, intrauterine distress or placental abruption before delivery; (2) asphyxia, resuscitation and rescue history, circulatory dysfunction and infection during or after delivery; and (3) early convulsions.

1.2 Assessment of brain injury MRI scans were analyzed by a radiologist and a newborn pediatrician who were unfamiliar with the clinical history. WMI diagnosis was carried out as described by reference, with some improvements.

1.3 Collection of clinical data Data, including delivery by cesarean section, gestational hypertension, diabetes mellitus, premature rupture of membranes and placental abruption, were collected for the mothers. Gestational age, weight, gender, whether small for gestational age, Apgar score, resuscitation history, circulatory disorders, early-onset sepsis, convulsions, and MRI data were collected for the newborns.

History of resuscitation and rescue refers to positive pressure ventilation, tracheal intubation, chest compression or epinephrine application during labor; circulatory disorders include at least two of the following indicators: prolonged capillary filling time, hypotension, oliguria, increased heart rate and increased liver.

1.4 Instrumentation MRI of the head was performed using an Intera Achieva 3.0T MRI system (Philips, Best, Netherlands). All infants were scanned by conventional MRI and diffusion-weighted imaging (DWI). Because of the retrospective study design, there are differences in imaging schemes, sequences and parameters measured.

ELIGIBILITY:
Inclusion Criteria:

* MRI head examination with informed consent of guardian
* Age 34-36+6 weeks

Exclusion Criteria:

* Other encephalopathies or congenital abnormality of brain development except white matter injury were excluded

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Late preterm infants undergoing head MRI, who were hospitalized in Shengjing Hospital from 1st January 2009 to 31st December 2022, were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2009-01; Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Imaging evaluation of different types of white matter injury in late preterm infants | 2009.1-2022.12
  The number of participants of white matter injury in late preterm infants, number of late preterm infants with different degrees (mild, moderate, severe) white matter injury and the imaging and pathological characteristics of early white matter injury (within 2 weeks after birth) using T1WI,T2WI,DWI,SWI.
Imaging differentiation of hemorrhagic and non hemorrhagic injuries | 2009.1-2022.12
  Using magnetic resonance technology, especially magnetic sensitivity, to identify and classify the cases of white matter injury in late preterm infants with or without hemorrhagic injury
Number of late preterm infants and distribution of gray matter injury in late preterm infants with white matter injury | 2009.1-2022.12
  Using magnetic resonance technology, To determine the number of gray matter injuries (cortex, thalamus, basal ganglia, brainstem) in late preterm infants with white matter injury
The number and distribution of PVL like injury in white matter injury of late preterm infants | 2009.1-2022.12
  Using magnetic resonance technology, to determine the probability of PVL-like injury in white matter injury of late preterm infants and which type and location are more prone to PVL-like outcomes

SECONDARY OUTCOMES:
Record of gestational age | 2009.1-2022.12
  To identify the high risk factors of brain white matter injury in late preterm infants，gestational age(weeks) of every late preterm infant will be recorded
Record of weight | 2009.1-2022.12
  To identify the high risk factors of brain white matter injury in late preterm infants，weight(g) of every late preterm infant will be recorded
Record of gender | 2009.1-2022.12
  To identify the high risk factors of brain white matter injury in late preterm infants， gender(male/female) of every late preterm infant will be recorded
Record of small for gestational age | 2009.1-2022.12
  To identify the high risk factors of brain white matter injury in late preterm infants，whether small for gestational age(yes/no) of every late preterm infant will be recorded
Record of apgar score | 2009.1-2022.12
  To identify the high risk factors of brain white matter injury in late preterm infants，Apgar score(1-10) of every late preterm infant will be recorded
Number of resuscitation history | 2009.1-2022.12
  To identify the high risk factors of brain white matter injury in late preterm infants，resuscitation history(yes/no) of every late preterm infant will be recorded.History of resuscitation and rescue refers to positive pressure ventilation, tracheal intubation, chest compression or epinephrine application during labor
Number of circulatory disorders | 2009.1-2022.12
  To identify the high risk factors of brain white matter injury in late preterm infants，circulatory disorders(yes/no) of every late preterm infant will be recorded.Circulatory disorders include at least two of the following indicators: prolonged capillary filling time, hypotension, oliguria, increased heart rate and increased liver.
Number of early-onset sepsis | 2009.1-2022.12
  To identify the high risk factors of brain white matter injury in late preterm infants，early-onset sepsis(yes/no) of every late preterm infant will be recorded
Number of convulsions | 2009.1-2022.12
  To identify the high risk factors of brain white matter injury in late preterm infants，convulsions(yes/no) of every late preterm infant will be recorded
Record of delivery by cesarean section | 2009.1-2022.12
  To identify the high risk factors of brain white matter injury in late preterm infants，delivery by cesarean section(yes/no) of every mother will be recorded
Number of gestational hypertension | 2009.1-2022.12
  To identify the high risk factors of brain white matter injury in late preterm infants，gestational hypertension(mmHg) of every mother will be recorded
Number of diabetes mellitus | 2009.1-2022.12
  To identify the high risk factors of brain white matter injury in late preterm infants，diabetes mellitus(yes/no) of every mother will be recorded
Number of premature rupture of membranes | 2009.1-2022.12
  To identify the high risk factors of brain white matter injury in late preterm infants，premature rupture of membranes(yes/no) of every mother will be recorded
Number of placental abruption | 2009.1-2022.12
  To identify the high risk factors of brain white matter injury in late preterm infants，placental abruption(yes/no) of every mother will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Jian Mao, doctor, Study Director — Shengjing Hospital
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No
Sharing the imaging results.

REFERENCES:
- [Result] Kinney HC. The near-term (late preterm) human brain and risk for periventricular leukomalacia: a review. Semin Perinatol. 2006 Apr;30(2):81-8. doi: 10.1053/j.semperi.2006.02.006. PMID 16731282
- [Result] Petrini JR, Dias T, McCormick MC, Massolo ML, Green NS, Escobar GJ. Increased risk of adverse neurological development for late preterm infants. J Pediatr. 2009 Feb;154(2):169-76. doi: 10.1016/j.jpeds.2008.08.020. Epub 2008 Dec 10. PMID 19081113
- [Result] Limperopoulos C, Soul JS, Gauvreau K, Huppi PS, Warfield SK, Bassan H, Robertson RL, Volpe JJ, du Plessis AJ. Late gestation cerebellar growth is rapid and impeded by premature birth. Pediatrics. 2005 Mar;115(3):688-95. doi: 10.1542/peds.2004-1169. PMID 15741373
- [Result] Guihard-Costa AM, Larroche JC. Differential growth between the fetal brain and its infratentorial part. Early Hum Dev. 1990 Jun;23(1):27-40. doi: 10.1016/0378-3782(90)90126-4. PMID 2209474
- [Result] Huppi PS, Warfield S, Kikinis R, Barnes PD, Zientara GP, Jolesz FA, Tsuji MK, Volpe JJ. Quantitative magnetic resonance imaging of brain development in premature and mature newborns. Ann Neurol. 1998 Feb;43(2):224-35. doi: 10.1002/ana.410430213. PMID 9485064
- [Result] Ballabh P, Braun A, Nedergaard M. Anatomic analysis of blood vessels in germinal matrix, cerebral cortex, and white matter in developing infants. Pediatr Res. 2004 Jul;56(1):117-24. doi: 10.1203/01.PDR.0000130472.30874.FF. Epub 2004 May 5. PMID 15128918
- [Result] Arrigoni F, Parazzini C, Righini A, Doneda C, Ramenghi LA, Lista G, Triulzi F. Deep medullary vein involvement in neonates with brain damage: an MR imaging study. AJNR Am J Neuroradiol. 2011 Dec;32(11):2030-6. doi: 10.3174/ajnr.A2687. Epub 2011 Sep 29. PMID 21960491
- [Result] Taoka T, Fukusumi A, Miyasaka T, Kawai H, Nakane T, Kichikawa K, Naganawa S. Structure of the Medullary Veins of the Cerebral Hemisphere and Related Disorders. Radiographics. 2017 Jan-Feb;37(1):281-297. doi: 10.1148/rg.2017160061. PMID 28076020
- [Result] Vilan A, Ribeiro JM, Reis C, Sampaio L. Deep Medullary Veins and Brain Injury. J Pediatr. 2018 Sep;200:290-290.e1. doi: 10.1016/j.jpeds.2018.03.051. Epub 2018 May 3. No abstract available. PMID 29731359
- [Result] du Plessis AJ. Cerebrovascular injury in premature infants: current understanding and challenges for future prevention. Clin Perinatol. 2008 Dec;35(4):609-41, v. doi: 10.1016/j.clp.2008.07.010. PMID 19026331
- [Result] Martinez-Biarge M, Groenendaal F, Kersbergen KJ, Benders MJ, Foti F, Cowan FM, de Vries LS. MRI Based Preterm White Matter Injury Classification: The Importance of Sequential Imaging in Determining Severity of Injury. PLoS One. 2016 Jun 3;11(6):e0156245. doi: 10.1371/journal.pone.0156245. eCollection 2016. PMID 27257863
- [Result] Ramenghi LA, Govaert P, Fumagalli M, Bassi L, Mosca F. Neonatal cerebral sinovenous thrombosis. Semin Fetal Neonatal Med. 2009 Oct;14(5):278-83. doi: 10.1016/j.siny.2009.07.010. Epub 2009 Aug 20. PMID 19699161
- [Result] Nakamura Y, Okudera T, Hashimoto T. Vascular architecture in white matter of neonates: its relationship to periventricular leukomalacia. J Neuropathol Exp Neurol. 1994 Nov;53(6):582-9. doi: 10.1097/00005072-199411000-00005. PMID 7964899
- [Result] Takashima S, Mito T, Ando Y. Pathogenesis of periventricular white matter hemorrhages in preterm infants. Brain Dev. 1986;8(1):25-30. doi: 10.1016/s0387-7604(86)80116-4. PMID 3486608
- [Result] Gould SJ, Howard S, Hope PL, Reynolds EO. Periventricular intraparenchymal cerebral haemorrhage in preterm infants: the role of venous infarction. J Pathol. 1987 Mar;151(3):197-202. doi: 10.1002/path.1711510307. PMID 3572613
- [Result] deVeber G, Andrew M, Adams C, Bjornson B, Booth F, Buckley DJ, Camfield CS, David M, Humphreys P, Langevin P, MacDonald EA, Gillett J, Meaney B, Shevell M, Sinclair DB, Yager J; Canadian Pediatric Ischemic Stroke Study Group. Cerebral sinovenous thrombosis in children. N Engl J Med. 2001 Aug 9;345(6):417-23. doi: 10.1056/NEJM200108093450604. PMID 11496852
- [Result] Moharir MD, Shroff M, Pontigon AM, Askalan R, Yau I, Macgregor D, Deveber GA. A prospective outcome study of neonatal cerebral sinovenous thrombosis. J Child Neurol. 2011 Sep;26(9):1137-44. doi: 10.1177/0883073811408094. Epub 2011 May 31. PMID 21628696
- [Result] Yang JY, Chan AK, Callen DJ, Paes BA. Neonatal cerebral sinovenous thrombosis: sifting the evidence for a diagnostic plan and treatment strategy. Pediatrics. 2010 Sep;126(3):e693-700. doi: 10.1542/peds.2010-1035. Epub 2010 Aug 9. PMID 20696732
- [Result] Doneda C, Righini A, Parazzini C, Arrigoni F, Rustico M, Triulzi F. Prenatal MR imaging detection of deep medullary vein involvement in fetal brain damage. AJNR Am J Neuroradiol. 2011 Sep;32(8):E146-9. doi: 10.3174/ajnr.A2249. Epub 2010 Oct 14. PMID 20947647
- [Result] Saxonhouse MA. Thrombosis in the Neonatal Intensive Care Unit. Clin Perinatol. 2015 Sep;42(3):651-73. doi: 10.1016/j.clp.2015.04.010. PMID 26250924
- [Result] Benninger KL, Maitre NL, Ruess L, Rusin JA. MR Imaging Scoring System for White Matter Injury after Deep Medullary Vein Thrombosis and Infarction in Neonates. AJNR Am J Neuroradiol. 2019 Feb;40(2):347-352. doi: 10.3174/ajnr.A5940. Epub 2019 Jan 17. PMID 30655251
- [Result] Pierson CR, Folkerth RD, Billiards SS, Trachtenberg FL, Drinkwater ME, Volpe JJ, Kinney HC. Gray matter injury associated with periventricular leukomalacia in the premature infant. Acta Neuropathol. 2007 Dec;114(6):619-31. doi: 10.1007/s00401-007-0295-5. Epub 2007 Oct 3. PMID 17912538